CLINICAL TRIAL: NCT02221037
Title: A Placebo Controlled, Double-blind, Multi-centre, Single Dose, Parallel Group, Randomised Clinical Trial of GSK2862277 in Patients Undergoing Oesophagectomy Surgery
Brief Title: Study of GSK2862277 in Subjects Undergoing Oesophagectomy Surgery
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated on the basis that protocol defined stopping criteria had been met.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 116341; 2014-000643-33 (EudraCT Number)
Record Dates: First submitted 2014-08-18; First posted 2014-08-20 (Estimated); Results first posted 2019-01-11 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Lung Injury, Acute and Respiratory Distress Syndrome, Adult
Keywords: PaO2/FiO2; Peri-operative lung injury; EVLWI; ARDS; PVPI; SOFA scores; GSK2862277; Oesophagectomy
MeSH Terms: conditions — Lung Injury; Respiratory Distress Syndrome | interventions — GSK2862277

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- GSK2862277 (Experimental): GSK2862277 will be administered as single orally inhaled aerosol over approximately 3 to 5 minutes; approximately 1-3 hours prior to the subjects scheduled surgery, before the initiation of pre-operative procedures. After surgery subject will undergo either ventilated or collapsed lung BAL procedure. Regular assessments will be conducted until the time of patient discharge. Subjects will be followed up as outpatients at Day 28
  Interventions: Drug: GSK2862277
- Placebo (Placebo Comparator): Placebo will be administered as single orally inhaled aerosol over approximately 3 to 5 minutes; approximately 1-3 hours prior to the subjects scheduled surgery, before the initiation of pre-operative procedures. After surgery subject will be undergo either ventilated or collapsed lung BAL procedure. Regular assessments will conducted until the time of patient discharge. Subjects will be followed up as outpatients at Day 28
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GSK2862277 — It is available as 26 milligrams (mg) white to off-white, uniform lyophilized cake that will be reconstituted (using reconstitution fluid formulated with polysorbate 80 in Water for Injection) to 40 mg/vial of Lyophile for reconstitution for inhalation with duration of nebulisation as approximately 3-5 min and will be administered using "Pari eFlow with s30 mesh" device.
  Arms: GSK2862277
Drug: Placebo — It is a clear, colorless to pale yellow liquid, will be administered in volume to match active dose as solution for inhalation with duration of nebulisation as approximately 3-5 min and will be administered using "Pari eFlow with s30 mesh" device.
  Arms: Placebo

SUMMARY:
Lung injury in patients undergoing oesophagectomy may occur during surgery (peri-operatively) as a result of One Lung Ventilation (OLV) and/or during the immediate post-operative period when patients receive intensive care. This is reinforced by the observation that physiological markers of lung injury are most elevated immediately after completion of surgery, and the development of clinical Acute Respiratory Distress Syndrome (ARDS)occurs immediately post-operatively (within 72 hours of surgery), with the majority of cases reported 24-48 hours after completion of surgery. This study is designed to investigate the impact of pre-operative administration of GSK2862277 on biological and physiological markers of lung injury in patients undergoing surgical resection of oesophageal cancer in order to achieve optimal exposure at the site of injury following OLV and lung deflation. This study is a randomized placebo controlled, double-blind, multi-centre, single dose parallel group, design. There will be two treatment groups comprising one active and one placebo arm with approximately 40 patients per group. Patients enrolled in the study will be scheduled to undergo planned/elective trans-thoracic surgery for oesophagectomy. The primary endpoint for this study is the change in pulmonary vascular permeability index (PVPI) from pre-surgical levels to the end of surgery. GSK2862277 will be administered as an orally inhaled aerosol (single nebulized dose) over approximately 3 to 5 minutes (min) 1-3 hours prior to surgery. Subject will be monitored daily until discharge and followed up till day 28.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a planned elective transthoracic oesophagectomy
* Male or female between 18 and 80 years of age inclusive, at the time of signing the informed consent.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* A female subject is eligible to participate if she is of:
* Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 milli-International Units per milliliter and estradiol < 40 picograms per milliliter (<147 picomoles per liter) is confirmatory]. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrolment. For most forms of HRT, at least 2-4 weeks should elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method.
* Liver parameters according to the thresholds below: Aspartate aminotransferase and Alanine aminotransferase < 5x Upper limit of normal (ULN); alkaline phosphatase and bilirubin <=1.5xULN (isolated bilirubin >1.5x ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* QT duration corrected for heart rate by Bazett's formula (QTcB) or QT duration corrected for heart rate by Fridericia's formula (QTcF) <= 480 milliseconds (msec) at screening
* Either QTcB or QTcF, machine or manual over-read can be used. This applies to both males and females. The QT correction formula used to determine inclusion and discontinuation for an individual subject should be the same throughout the study.
* Based on average QTc value of triplicate ECGs obtained over a brief recording period.

Exclusion Criteria:

* Positive screening test for pre-existing antibodies that bind GSK2862277.
* Current evidence or history of pneumonia within 14 days before dosing.
* Diagnosis of chronic respiratory disease with a forced expiratory volume in one second (FEV1) less than 50% predicted or resting oxygen saturations of less 92%.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* The subject has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Use of corticosteroids (Intravenous, oral or Intramuscular) at a dose of >= 10 Milligrams per day (mg/day) prednisolone (or equivalent) within 14 days prior to dosing, or anti-Tumor Necrosis Factor (anti-TNF) or anti-IL1 within 60 days prior to dosing.

Criteria Based Upon Medical Histories

* History or current evidence of clinically significant renal disease, diabetes mellitus/metabolic syndrome, hypertension, peripheral vascular disease or any other clinically significant respiratory, cardiovascular, neurological, endocrine, or hematological abnormalities that are uncontrolled on permitted therapy. Significant is defined as any disease that, in the opinion of the Investigator, would put the safety of the patients at risk through study participation, or which would affect the safety analysis or other analysis if the disease/condition exacerbated during the study.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* History of regular alcohol consumption within 6 months of the study, defined as: an average weekly intake of >28 units for males or >14 units for females. One unit is equivalent to 8 grams of alcohol: a half-pint [~240 milliliter (ml)] of beer, 1 glass (125 ml) of wine or 1 (25 ml) measure of spirits Criteria Based Upon Diagnostic Assessments
* Screens positive for Hepatitis B surface antigen, Hepatitis C antibody
* Known Human Immunodeficiency Virus (HIV) positive; testing will be conducted in accordance with local procedures
* Tests positive for Mycobacterium tuberculosis using QuantiFERON Gold Test. Other Criteria
* Subject has received a live attenuated vaccine(s) within 3 weeks of randomisation or will require vaccination with a live attenuated vaccine prior to the end of the study (Day 28).
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subject is mentally or legally incapacitated.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2015-04-28 (Actual); Primary Completion 2017-06-28 (Actual); Study Completion 2017-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (5):
- United Kingdom (5):
  - GSK Investigational Site, Cottingham, Yorkshire
  - GSK Investigational Site, Belfast
  - GSK Investigational Site, Birmingham
  - GSK Investigational Site, Cambridge
  - GSK Investigational Site, Middlesbrough

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study is available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (copy the URL below to your browser)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://www.clinicalstudydatarequest.com/Posting.aspx?ID=20588

REFERENCES:
- [Background] Ryan J, Bayliffe AI, McAuley DF, Yeung J, Thickett DR, Howells PA, O'Donnell C, Vassallo AM, Wright TJ, McKie E, Hardes K, Summers C, Shields MO, Powley W, Wilson R, Lazaar AL, Fowler A, Perkins GD. A nebulised antitumour necrosis factor receptor-1 domain antibody in patients at risk of postoperative lung injury: A randomised, placebo-controlled pilot study. Eur J Anaesthesiol. 2020 Nov;37(11):1014-1024. doi: 10.1097/EJA.0000000000001245. PMID 32467417

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 8 centers in the United Kingdom from 28-Apr-2015 to 28-Jun-2017.
Pre-assignment Details: A total of 54 participants (included 2 participants who were screen-failures and were re-screened) were screened, of which 21 participants (2 re-entered study) were screen-failures (SF). Reasons for SF: study procedure could not be performed (4), inclusion/exclusion criteria not met (14), study closed/terminated (1) and investigator discretion (2).
Groups:
- Placebo (BAL Collapsed Lung): Eligible participants received a single dose of matching placebo on Day 1 via oral inhalation route over approximately 3 to 5 minutes; approximately 1 to 3 hours prior to scheduled surgery. After surgery, participants in this arm underwent collapsed lung broncho-alveolar lavage (BAL) procedure on Day 1.
- Placebo (BAL Ventilated Lung): Eligible participants received a single dose of matching placebo on Day 1 via oral inhalation route over approximately 3 to 5 minutes; approximately 1 to 3 hours prior to scheduled surgery. After surgery, participants in this arm underwent ventilated lung BAL procedure on Day 1.
- GSK2862277 26 mg (BAL Collapsed Lung): Eligible participants received a single dose of GSK2862277 26 milligrams (mg) on Day 1 via oral inhalation route over approximately 3 to 5 minutes; approximately 1 to 3 hours prior to scheduled surgery. After surgery, participants in this arm underwent collapsed lung BAL procedure on Day 1.
- GSK2862277 26 mg (BAL Ventilated Lung): Eligible participants received a single dose of GSK2862277 26 mg on Day 1 via oral inhalation route over approximately 3 to 5 minutes; approximately 1 to 3 hours prior to scheduled surgery. After surgery, participants in this arm underwent ventilated lung BAL procedure on Day 1.
Period: Overall Study
Arm/Group | Placebo (BAL Collapsed Lung) | Placebo (BAL Ventilated Lung) | GSK2862277 26 mg (BAL Collapsed Lung) | GSK2862277 26 mg (BAL Ventilated Lung)
Started | 5 | 11 | 8 | 9
Completed | 5 | 11 | 7 | 9
Not Completed | 0 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population which comprised of all participants who received at least one complete dose of study treatment.
Groups:
- Placebo (BAL Collapsed Lung): Eligible participants received a single dose of matching placebo on Day 1 via oral inhalation route over approximately 3 to 5 minutes; approximately 1 to 3 hours prior to scheduled surgery. After surgery, participants in this arm underwent collapsed lung BAL procedure on Day 1.
- GSK2862277 26 mg (BAL Collapsed Lung): Eligible participants received a single dose of GSK2862277 26 mg on Day 1 via oral inhalation route over approximately 3 to 5 minutes; approximately 1 to 3 hours prior to scheduled surgery. After surgery, participants in this arm underwent collapsed lung BAL procedure on Day 1.
- Total: Total of all reporting groups
Arm/Group | Placebo (BAL Collapsed Lung) | Placebo (BAL Ventilated Lung) | GSK2862277 26 mg (BAL Collapsed Lung) | GSK2862277 26 mg (BAL Ventilated Lung) | Total
Number analyzed (Participants) | 5 | 11 | 8 | 9 | 33
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.0 (9.70) | 63.5 (10.47) | 62.0 (4.69) | 59.3 (10.76) | 61.9 (9.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 4 | 0 | 2 | 6
  Male | 5 | 7 | 8 | 7 | 27
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 5 | 11 | 8 | 9 | 33

OUTCOME MEASURES:

1. Primary Outcome: Baseline Adjusted Change in Pulmonary Vascular Permeability Index (PVPI) on Completion of Surgery
Description: PVPI is a derived value from extra vascular lung water (EVLW), and is considered to be less variable than extra vascular lung water Index (EVLWI). PVPI was measured via single-indicator transpulmonary thermodilution with a patent indwelling Pulse Contour Cardiac Output (PiCCO) catheter. Baseline was Day 1 (immediately prior to start of surgery). Change from Baseline value was the post-Baseline value (on completion of surgery on Day 1) minus Baseline value. Per-Protocol 1 (PP1) Population comprised of all the participants in the Safety population for whom the treatment actually received was the same one when they were randomized to (both study drug and BAL sampling location).
Time Frame: Baseline (Day 1 [immediately prior to start of surgery]) and Day 1 (on completion of surgery)
Population: PP1 Population.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Placebo (BAL Collapsed Lung) | Placebo (BAL Ventilated Lung) | GSK2862277 26 mg (BAL Collapsed Lung) | GSK2862277 26 mg (BAL Ventilated Lung)
Number analyzed (Participants) | 5 | 10 | 5 | 8
Ratio | 0.00 (0.367) | 0.11 (0.664) | -0.18 (0.536) | 0.21 (0.449)

2. Secondary Outcome: Baseline Adjusted Change in EVLWI on Completion of Surgery
Description: EVLW refers to the fluid within the lung but outside the vascular compartment. It includes extravasated plasma, intracellular water, lymphatic fluid, and surfactant. EVLWI was measured by trans-pulmonary thermodilution via a PiCCO hemodynamic monitor. Baseline was Day 1 (immediately prior to start of surgery). Change from Baseline value was the post-Baseline value (on completion of surgery on Day 1) minus Baseline value. Only those participants with data available at the specified time points were analyzed.
Time Frame: Baseline (Day 1 [immediately prior to start of surgery]) and Day 1 (on completion of surgery)
Population: PP1 Population.
Measure: Mean (Standard Deviation); unit: Milliliters per kilograms
Arm/Group | Placebo (BAL Collapsed Lung) | Placebo (BAL Ventilated Lung) | GSK2862277 26 mg (BAL Collapsed Lung) | GSK2862277 26 mg (BAL Ventilated Lung)
Number analyzed (Participants) | 5 | 8 | 5 | 8
Milliliters per kilograms | 0.462 (1.4731) | -0.317 (1.3436) | 0.008 (1.2527) | -0.300 (3.8403)

3. Secondary Outcome: Number of Participants With Adverse Events (AE) and Serious Adverse Events (SAE)
Description: AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with use of a medicinal product (MP), whether or not considered related to MP. AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with use of MP. SAE is any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect or is medically significant or all events of possible drug induced liver injury with hyperbilirubinemia. Safety Population comprised of all participants who received at least one complete dose of study treatment.
Time Frame: Up to Day 31
Population: Safety Population.
Measure: Number; unit: Participants
Arm/Group | Placebo (BAL Collapsed Lung) | Placebo (BAL Ventilated Lung) | GSK2862277 26 mg (BAL Collapsed Lung) | GSK2862277 26 mg (BAL Ventilated Lung)
Number analyzed (Participants) | 5 | 11 | 8 | 9
Participants
  AE | 5 | 10 | 6 | 9
  SAE | 3 | 5 | 5 | 4

4. Secondary Outcome: Number of Participants With Hematology Abnormalities of Potential Clinical Importance
Description: Hematology parameters included basophils, eosinophils, hematocrit, hemoglobin, lymphocytes, monocytes, neutrophils, neutrophil bands, platelets, red blood cell (RBC) count, segmented neutrophils and white blood cell (WBC) count. The potential clinical concern values were: hematocrit (low: <0.3 fraction and high: >0.54 fraction), Hemoglobin (low: <90 gram per Liter and high: >180 gram per Liter), lymphocytes (low: <0.6 x 10^9 cells/Liter and high: >3.0 x 10^9 cells/Liter), neutrophils: (low: <1.5 x 10^9 cells/Liter and high: >20 x 10^9 cells/Liter), platelets: (low: <100 x 10^9 cells/Liter and high: >600 x 10^9 cells/Liter) and WBC: (low: <3 x 10^9 cells/Liter and high: >20 x 10^9 cells/Liter). Only those participants for which at least one value of potential clinical concern was reported are summarized.
Time Frame: Up to Day 8
Population: Safety Population.
Measure: Number; unit: Participants
Arm/Group | Placebo (BAL Collapsed Lung) | Placebo (BAL Ventilated Lung) | GSK2862277 26 mg (BAL Collapsed Lung) | GSK2862277 26 mg (BAL Ventilated Lung)
Number analyzed (Participants) | 5 | 11 | 8 | 9
Participants | 5 | 10 | 5 | 8

5. Secondary Outcome: Number of Participants With Clinical Chemistry Abnormalities of Potential Clinical Importance
Description: Clinical chemistry parameters and their potential clinical concern values were: albumin (low: <25 millimole [mmol]/L and high: >60 mmol/L), calcium (low: <1.8 mmoL/L and high: >2.75 mmol/L), creatinine (low: <30 mmol/L and high: >160 mmol/L), glucose (low: <3 mmol/L and high: >9 mmol/L), potassium (low: <2.5 mmol/L and high: >5.5 mmol/L), sodium (low: <120 mmol/L and high: >160 mmol/L), total carbon dioxide content (low: <16 mmol/L and high: >35 mmol/L) and blood urea nitrogen (low: <3 mmol/L and high: >15 mmol/L). Number of participants with clinical chemistry abnormalities of potential clinical importance are presented.
Time Frame: Up to Day 8
Population: Safety Population.
Measure: Number; unit: Participants
Arm/Group | Placebo (BAL Collapsed Lung) | Placebo (BAL Ventilated Lung) | GSK2862277 26 mg (BAL Collapsed Lung) | GSK2862277 26 mg (BAL Ventilated Lung)
Number analyzed (Participants) | 5 | 11 | 8 | 9
Participants | 4 | 5 | 4 | 4

6. Secondary Outcome: Number of Participants With Abnormal Urinalysis Parameters
Description: Urinalysis included dipstick urine test which was used to screen for glucose, ketones, occult blood and protein on Day 1 (pre-dose) and Day 8. The dipstick test gives results in a semi-quantitative manner, and results for urinalysis parameters of urine glucose, ketones, occult blood and protein can be read as Trace, 1+, 2+ and 3+, indicating proportional concentrations in the urine sample.
Time Frame: Day 1 (pre-dose) and Day 8
Population: Safety Population.
Measure: Number; unit: Participants
Arm/Group | Placebo (BAL Collapsed Lung) | Placebo (BAL Ventilated Lung) | GSK2862277 26 mg (BAL Collapsed Lung) | GSK2862277 26 mg (BAL Ventilated Lung)
Number analyzed (Participants) | 5 | 11 | 8 | 9
Participants
  Urine glucose: Day 1 (pre-dose): Trace | 0 | 0 | 0 | 0
  Urine glucose: Day 1 (pre-dose): 1+ | 0 | 0 | 0 | 0
  Urine glucose: Day 1 (pre-dose): 2+ | 1 | 0 | 0 | 0
  Urine glucose: Day 1 (pre-dose): 3+ | 0 | 0 | 1 | 0
  Urine glucose: Day 8: Trace | 0 | 1 | 0 | 2
  Urine glucose: Day 8: 1+ | 0 | 0 | 0 | 0
  Urine glucose: Day 8: 2+ | 1 | 0 | 0 | 0
  Urine glucose: Day 8: 3+ | 0 | 0 | 0 | 0
  Urine ketones: Day 1 (pre-dose): Trace | 1 | 0 | 1 | 0
  Urine ketones: Day 1 (pre-dose): 1+ | 0 | 0 | 0 | 0
  Urine ketones: Day 1 (pre-dose): 2+ | 0 | 0 | 0 | 0
  Urine ketones: Day 1 (pre-dose): 3+ | 0 | 0 | 0 | 0
  Urine ketones: Day 8: Trace | 0 | 0 | 0 | 2
  Urine ketones: Day 8: 1+ | 0 | 0 | 1 | 0
  Urine ketones: Day 8: 2+ | 0 | 0 | 0 | 0
  Urine ketones: Day 8: 3+ | 0 | 0 | 0 | 0
  Urine occult blood: Day 1 (pre-dose): Trace | 0 | 0 | 1 | 0
  Urine occult blood: Day 1 (pre-dose): 1+ | 0 | 2 | 1 | 0
  Urine occult blood: Day 1 (pre-dose): 2+ | 0 | 0 | 0 | 0
  Urine occult blood: Day 1 (pre-dose): 3+ | 0 | 0 | 0 | 0
  Urine occult blood: Day 8: Trace | 0 | 0 | 0 | 0
  Urine occult blood: Day 8: 1+ | 1 | 1 | 0 | 0
  Urine occult blood: Day 8: 2+ | 0 | 0 | 0 | 2
  Urine occult blood: Day 8: 3+ | 0 | 1 | 0 | 0
  Urine protein: Day 1 (pre-dose): Trace | 0 | 0 | 0 | 2
  Urine protein: Day 1 (pre-dose): 1+ | 1 | 0 | 1 | 0
  Urine protein: Day 1 (pre-dose): 2+ | 0 | 1 | 0 | 1
  Urine protein: Day 1 (pre-dose): 3+ | 0 | 0 | 0 | 0
  Urine protein: Day 8: Trace | 1 | 5 | 0 | 3
  Urine protein: Day 8: 1+ | 2 | 4 | 2 | 2
  Urine protein: Day 8: 2+ | 0 | 0 | 1 | 2
  Urine protein: Day 8: 3+ | 0 | 0 | 0 | 0

7. Secondary Outcome: Number of Participants With Electrocardiogram (ECG) Values of Potential Clinical Importance
Description: Single 12-lead ECGs were obtained thereafter during the study, using an ECG machine that automatically calculated the heart rate and measured PR, QRS, QT, RR and corrected QT (QTc) intervals. Number of participants with ECG values of potential clinical importance are presented.
Time Frame: Days 1, 2, 4 and 8
Population: Safety Population.
Measure: Number; unit: Participants
Arm/Group | Placebo (BAL Collapsed Lung) | Placebo (BAL Ventilated Lung) | GSK2862277 26 mg (BAL Collapsed Lung) | GSK2862277 26 mg (BAL Ventilated Lung)
Number analyzed (Participants) | 5 | 11 | 8 | 9
Participants | 5 | 7 | 4 | 8

8. Secondary Outcome: Number of Participants With Vital Signs of Potential Clinical Importance
Description: Vital sign measurements included systolic and diastolic blood pressure, pulse rate, temperature and respiratory rate. Vital sign measurements were measured in a semi-recumbent or supine position after 5 minutes rest. The potential clinical concern range for systolic blood pressure: <85 and >160 millimeters of mercury, for diastolic: <45 and >100 millimeters of mercury and heart rate: <40 and >110 beats per minute. Number of participants with vital signs of potential clinical importance are presented.
Time Frame: Up to Day 31
Population: Safety Population.
Measure: Number; unit: Participants
Arm/Group | Placebo (BAL Collapsed Lung) | Placebo (BAL Ventilated Lung) | GSK2862277 26 mg (BAL Collapsed Lung) | GSK2862277 26 mg (BAL Ventilated Lung)
Number analyzed (Participants) | 5 | 11 | 8 | 9
Participants | 2 | 3 | 3 | 3

9. Secondary Outcome: Baseline Adjusted Change in PaO2/FiO2 on Completion of Surgery
Description: Oxygenation and function of gas exchange was assessed by the comparison of partial pressure of oxygen arterially (PaO2) divided by the fraction of oxygen that is being inspired (FiO2), sometimes referred to simply as the 'P to F ratio'. The P to F ratio was assessed at time points during the period of intubation and mechanical ventilation. An arterial blood sample was required for determination of the partial pressure of oxygen and the percentage of O2 which is being inspired was recorded at the corresponding time point. Baseline was Day 1 (immediately prior to start of surgery). Change from Baseline value was the post-Baseline value (on completion of surgery on Day 1) minus Baseline value.
Time Frame: Baseline (Day 1 [immediately prior to start of surgery]) and Day 1 (on completion of surgery)
Population: PP1 Population.
Measure: Mean (Standard Deviation); unit: Millimiters of Mercury
Arm/Group | Placebo (BAL Collapsed Lung) | Placebo (BAL Ventilated Lung) | GSK2862277 26 mg (BAL Collapsed Lung) | GSK2862277 26 mg (BAL Ventilated Lung)
Number analyzed (Participants) | 5 | 10 | 5 | 8
Millimiters of Mercury | 8.9 (141.10) | 18.5 (160.82) | -47.5 (252.16) | 11.2 (98.12)

10. Secondary Outcome: Levels of BAL Biomarkers on Completion of Surgery
Description: Samples were collected to determine concentrations of biomarkers in BAL using an appropriately validated assay on Day 1 after completion of surgery. BAL biomarkers included soluble tumor necrosis factor receptor (STNFR) type I, free, STNFR type I, total, tumor necrosis factor alpha, interleukin 6, interleukin 8, interleukin 1 beta, monocyte chemotactic protein-1, macrophage inflammatory protein 1 alpha, macrophage inflammatory protein 1 beta, interleukin 10 and soluble receptor for advanced glycation end (sRAGE) products. Any value below limit of quantification was replaced with half the lower limit of quantification (LLQ) prior to deriving the summary measures. Mean levels of BAL biomarkers on completion of surgery are presented. Only those participants available at the specified time points were analyzed represented by n=X,X,X,X in the category titles.
Time Frame: Day 1 (on completion of surgery)
Population: PP1 Population.
Measure: Mean (Standard Deviation); unit: Picograms per milliliter
Arm/Group | Placebo (BAL Collapsed Lung) | Placebo (BAL Ventilated Lung) | GSK2862277 26 mg (BAL Collapsed Lung) | GSK2862277 26 mg (BAL Ventilated Lung)
Number analyzed (Participants) | 5 | 10 | 5 | 8
Picograms per milliliter
  STNFR type I, Free, n=5,9,5,8: number analyzed (Participants) | 5 | 9 | 5 | 8
  STNFR type I, Free, n=5,9,5,8 | 645.5400 (398.14834) | 278.2529 (201.58668) | 106.1600 (168.39828) | 67.7713 (69.69634)
  STNFR I, Total, n=5,9,5,8: number analyzed (Participants) | 5 | 9 | 5 | 8
  STNFR I, Total, n=5,9,5,8 | 299.4000 (168.92556) | 310.8136 (307.29751) | 175.5660 (167.67312) | 183.9000 (229.72939)
  Tumor necrosis factor alpha, n=5,9,5,7: number analyzed (Participants) | 5 | 9 | 5 | 7
  Tumor necrosis factor alpha, n=5,9,5,7 | 3.5110 (2.68376) | 24.3850 (33.67945) | 6.1040 (12.51974) | 3.7814 (5.33211)
  Interleukin 6, n=5,9,5,8: number analyzed (Participants) | 5 | 9 | 5 | 8
  Interleukin 6, n=5,9,5,8 | 63.580 (66.8285) | 138.917 (217.3948) | 15.844 (30.5243) | 43.828 (64.0092)
  Interleukin 8, n=5,9,5,8: number analyzed (Participants) | 5 | 9 | 5 | 8
  Interleukin 8, n=5,9,5,8 | 8041.600 (16369.4998) | 3822.170 (6270.8199) | 126.340 (145.1019) | 432.513 (731.0601)
  Interleukin 1 beta, n=5,9,5,8: number analyzed (Participants) | 5 | 9 | 5 | 8
  Interleukin 1 beta, n=5,9,5,8 | 70.2376 (123.55622) | 66.3749 (99.46797) | 1.1674 (0.78732) | 18.6054 (38.61022)
  Monocyte chemotactic protein-1, n=5,9,5,8: number analyzed (Participants) | 5 | 9 | 5 | 8
  Monocyte chemotactic protein-1, n=5,9,5,8 | 118.1600 (124.52553) | 122.2649 (170.65326) | 53.4260 (75.21106) | 51.5713 (59.72512)
  Macrophage inflammatory protein 1 alpha, n=5,9,5,8: number analyzed (Participants) | 5 | 9 | 5 | 8
  Macrophage inflammatory protein 1 alpha, n=5,9,5,8 | 63.348 (54.8461) | 165.300 (203.2446) | 9.140 (0.0000) | 23.942 (32.7837)
  Macrophage inflammatory protein 1 beta, n=5,9,5,8: number analyzed (Participants) | 5 | 9 | 5 | 8
  Macrophage inflammatory protein 1 beta, n=5,9,5,8 | 142.040 (132.7086) | 219.891 (264.1694) | 28.292 (41.4424) | 48.413 (82.2684)
  Interleukin 10, n=5,9,5,8: number analyzed (Participants) | 5 | 9 | 5 | 8
  Interleukin 10, n=5,9,5,8 | 1.7098 (1.93498) | 5.2672 (8.39023) | 0.5130 (0.00000) | 1.8123 (3.23279)
  sRAGE products, n=5,9,5,8: number analyzed (Participants) | 5 | 9 | 5 | 8
  sRAGE products, n=5,9,5,8 | 1440.2 (1144.89) | 2121.7 (2078.47) | 1966.0 (2734.60) | 1044.6 (1560.45)

11. Secondary Outcome: Levels of BAL Biomarkers (C-reactive Protein and Total Proteins) on Completion of Surgery
Description: Samples were collected to determine concentrations of biomarkers in BAL using an appropriately validated assay. BAL biomarkers included C-reactive protein and total proteins. Any value below limit of quantification was replaced with half the LLQ prior to deriving the summary measures. All BAL C-reactive protein samples were below limit of quantification and all were assigned to half the LLQ prior to deriving the summary measures. Mean levels of BAL biomarkers on completion of surgery are presented. Only those participants available at the specified time points were analyzed represented by n=X,X,X,X in the category titles.
Time Frame: Day 1 (on completion of surgery)
Population: PP1 Population.
Measure: Mean (Standard Deviation); unit: Milligrams per Liter
Arm/Group | Placebo (BAL Collapsed Lung) | Placebo (BAL Ventilated Lung) | GSK2862277 26 mg (BAL Collapsed Lung) | GSK2862277 26 mg (BAL Ventilated Lung)
Number analyzed (Participants) | 5 | 10 | 5 | 8
Milligrams per Liter
  C-reactive protein, n=5,9,5,8: number analyzed (Participants) | 5 | 9 | 5 | 8
  C-reactive protein, n=5,9,5,8 | 0.04650 (0.000000) | 0.04650 (0.000000) | 0.04650 (0.000000) | 0.04650 (0.000000)
  Total proteins, n=5,10,5,8 | 423.6 (182.80) | 605.1 (670.60) | 136.8 (108.33) | 303.0 (274.85)

12. Secondary Outcome: Levels of BAL Biomarkers (Surfactant Protein and Clara Cell Secretory Protein) on Completion of Surgery
Description: Samples were collected to determine concentrations of biomarkers in BAL using an appropriately validated assay. BAL biomarkers included surfactant protein D and clara cell secretory protein. Any value below limit of quantification was replaced with half the LLQ prior to deriving the summary measures. Mean levels of BAL biomarkers on completion of surgery are presented. Only those participants available at the specified time points were analyzed represented by n=X,X,X,X in the category titles.
Time Frame: Day 1 (on completion of surgery)
Population: PP1 Population.
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter
Arm/Group | Placebo (BAL Collapsed Lung) | Placebo (BAL Ventilated Lung) | GSK2862277 26 mg (BAL Collapsed Lung) | GSK2862277 26 mg (BAL Ventilated Lung)
Number analyzed (Participants) | 5 | 10 | 5 | 8
Nanograms per milliliter
  Surfactant Protein D, n=5,9,5,8: number analyzed (Participants) | 5 | 9 | 5 | 8
  Surfactant Protein D, n=5,9,5,8 | 411.92 (472.487) | 760.04 (898.224) | 872.88 (848.358) | 551.31 (943.640)
  Clara cell secretory protein, n=5,7,5,7: number analyzed (Participants) | 5 | 7 | 5 | 7
  Clara cell secretory protein, n=5,7,5,7 | 3635.40 (2575.875) | 2131.66 (3217.852) | 1000.40 (1167.704) | 1409.21 (2358.501)

13. Secondary Outcome: Change Over Time in PaO2/FiO2 Post-operatively on Day 2 Through to Day 4
Description: Oxygenation and function of gas exchange was assessed by the comparison of PaO2 divided by the FiO2, sometimes referred to simply as the 'P to F ratio'. The P to F ratio was assessed at time points during the period of intubation and mechanical ventilation. An arterial blood sample was required for determination of the partial pressure of oxygen and the percentage of O2 which is being inspired was recorded at the corresponding time point. Baseline was Day 1 (immediately prior to start of surgery). Change from Baseline value was the post-Baseline value (on completion of surgery on Day 1) minus Baseline value. PP1 Population was analyzed. Only those participants available at the specified time points were analyzed represented by n=X,X in the category titles.
Time Frame: Baseline (Day 1 [immediately prior to start of surgery]) to Days 2, 3 and 4
Population: PP1 Population.
Measure: Mean (Standard Deviation); unit: Millimeters of Mercury
Arm/Group | Placebo (BAL Collapsed Lung) | Placebo (BAL Ventilated Lung) | GSK2862277 26 mg (BAL Collapsed Lung) | GSK2862277 26 mg (BAL Ventilated Lung)
Number analyzed (Participants) | 5 | 10 | 5 | 8
Millimeters of Mercury
  Day 2, n=5,8,5,6: number analyzed (Participants) | 5 | 8 | 5 | 6
  Day 2, n=5,8,5,6 | -15.1 (171.84) | -103.3 (87.24) | 38.9 (312.28) | -79.3 (199.85)
  Day 3, n=5,8,5,5: number analyzed (Participants) | 5 | 8 | 5 | 5
  Day 3, n=5,8,5,5 | -53.7 (120.35) | -43.0 (179.64) | -9.5 (325.46) | -119.0 (148.67)
  Day 4, n=5,8,5,5: number analyzed (Participants) | 5 | 8 | 5 | 5
  Day 4, n=5,8,5,5 | -36.3 (139.18) | -123.6 (68.14) | -22.3 (342.46) | -56.5 (123.31)

14. Secondary Outcome: Change Over Time in PVPI Post-operatively on Day 2 Through to Day 4
Description: PVPI is a derived value from EVLW, and is considered to be less variable than EVLWI. PVPI was measured via single-indicator transpulmonary thermodilution as long as the participant remained in the ICU with a patent indwelling PiCCO catheter. Baseline was Day 1 (immediately prior to start of surgery). Change from Baseline value was the post-Baseline value minus Baseline value. PP1 Population was analyzed. Only those participants available at the specified time points were analyzed represented by n=X,X,X,X in the category titles.
Time Frame: Baseline (Day 1 [immediately prior to start of surgery]) to Days 2, 3 and 4
Population: PP1 Population.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Placebo (BAL Collapsed Lung) | Placebo (BAL Ventilated Lung) | GSK2862277 26 mg (BAL Collapsed Lung) | GSK2862277 26 mg (BAL Ventilated Lung)
Number analyzed (Participants) | 5 | 10 | 5 | 8
Ratio
  Day 2, n=5,6,3,5: number analyzed (Participants) | 5 | 6 | 3 | 5
  Day 2, n=5,6,3,5 | -0.22 (0.259) | -0.27 (0.427) | -0.50 (0.346) | -0.42 (0.630)
  Day 3, n=4,6,3,5: number analyzed (Participants) | 4 | 6 | 3 | 5
  Day 3, n=4,6,3,5 | -0.20 (0.648) | -0.23 (0.516) | -0.30 (0.529) | -0.32 (0.756)
  Day 4, n=3,5,2,4: number analyzed (Participants) | 3 | 5 | 2 | 4
  Day 4, n=3,5,2,4 | -0.40 (0.200) | -0.24 (0.666) | -0.20 (0.000) | -0.08 (0.850)

15. Secondary Outcome: Change Over Time in EVLWI Post-operatively on Day 2 Through to Day 4
Description: EVLW refers to the fluid within the lung but outside the vascular compartment. It includes extravasated plasma, intracellular water, lymphatic fluid, and surfactant. EVLWI was measured by trans-pulmonary thermodilution via a PiCCO hemodynamic monitor. Change from Baseline value was the post-Baseline value minus Baseline value. PP1 Population was analyzed. Only those participants available at the specified time points were analyzed represented by n=X,X,X,X in the category titles.
Time Frame: Baseline (Day 1 [immediately prior to start of surgery]) to Days 2, 3 and 4
Population: PP1 Population.
Measure: Mean (Standard Deviation); unit: Millimeters per kilograms
Arm/Group | Placebo (BAL Collapsed Lung) | Placebo (BAL Ventilated Lung) | GSK2862277 26 mg (BAL Collapsed Lung) | GSK2862277 26 mg (BAL Ventilated Lung)
Number analyzed (Participants) | 5 | 10 | 5 | 8
Millimeters per kilograms
  Day 2, n=5,6,3,5: number analyzed (Participants) | 5 | 6 | 3 | 5
  Day 2, n=5,6,3,5 | -0.033 (1.1203) | -1.120 (2.4825) | -0.694 (0.8710) | 0.604 (1.3370)
  Day 3, n=4,5,3,5: number analyzed (Participants) | 4 | 5 | 3 | 5
  Day 3, n=4,5,3,5 | 0.062 (1.2468) | -0.190 (1.4762) | -0.203 (2.3349) | 0.755 (1.4801)
  Day 4, n=3,5,2,4: number analyzed (Participants) | 3 | 5 | 2 | 4
  Day 4, n=3,5,2,4 | -0.621 (0.2646) | 0.828 (4.1772) | 0.311 (1.9297) | 1.981 (2.8449)

16. Secondary Outcome: Daily Sequential Organ Failure Assessment (SOFA) Scores on Day 2 Through to Day 4
Description: The SOFA score defines the presence and severity of dysfunction within 6 organ systems (cardiovascular, respiratory, coagulation, liver, renal, and nervous system) with a value of "0" for assigned to normal function to a maximum value of "4" for severe dysfunction in each of the organ systems. Each component of the SOFA score was added together, ranging from "0" indicating no organ dysfunction in any of the 6 organ systems, to "24" indicating maximal organ dysfunction across all 6 organ systems. Per-Protocol (PP) 2 Population comprised of all the participants in the Safety population for whom the study drug actually received was the same one they were randomized to (study drug).
Time Frame: Day 2 to Day 4
Population: PP 2 Population.
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Placebo (BAL Collapsed Lung) | Placebo (BAL Ventilated Lung) | GSK2862277 26 mg (BAL Collapsed Lung) | GSK2862277 26 mg (BAL Ventilated Lung)
Number analyzed (Participants) | 5 | 11 | 6 | 8
Scores on a Scale
  Day 2 | 1.0 (2.24) | 1.6 (1.39) | 1.5 (2.54) | 2.1 (1.92)
  Day 3 | 3.4 (4.72) | 1.5 (1.80) | 1.8 (2.86) | 1.6 (1.43)
  Day 4 | 2.2 (3.96) | 1.3 (0.90) | 1.3 (3.56) | 1.6 (1.69)

17. Secondary Outcome: Area Under the Concentration-time Curve From Time Zero (Pre-dose) to Last Time of Quantifiable Concentration (AUC [0 to t])
Description: Blood samples for pharmacokinetic analysis of GSK2862277 were collected at the indicated time points. Pharmacokinetic (PK) Population comprised of all participants in the Safety population for whom a pharmacokinetic sample (plasma and/or BAL) was obtained and analyzed.
Time Frame: Day 1 (pre-dose, 1 hour post-dose and on completion of surgery), Day 2 (24 to 26 hours post-dose) and Day 3 (46 to 50 hours post-dose)
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*picograms/milliliter
Arm/Group | GSK2862277 26 mg (BAL Collapsed Lung) | GSK2862277 26 mg (BAL Ventilated Lung)
Number analyzed (Participants) | 3 | 6
Hours*picograms/milliliter | 340505.15 (45.284) | 290102.64 (76.450)

18. Secondary Outcome: Maximum Observed Concentration (Cmax)
Description: Blood samples for pharmacokinetic analysis of GSK2862277 were collected at the indicated time points.
Time Frame: as for outcome 17
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picograms per milliliters
Arm/Group | GSK2862277 26 mg (BAL Collapsed Lung) | GSK2862277 26 mg (BAL Ventilated Lung)
Number analyzed (Participants) | 3 | 6
Picograms per milliliters | 31123.58 (64.452) | 25469.14 (93.307)

19. Secondary Outcome: Derived Pharmacokinetic Parameter- Half-life (t1/2) and Time of Occurrence of Cmax (Tmax)
Description: Half-life (t1⁄2) is the time required for a quantity to reduce to half its initial value. t1/2 was not determined in all cases due to insufficient data in the terminal phase. Blood samples for pharmacokinetic analysis of GSK2862277 were collected at the indicated time points. Only those participants available at the specified time points were analyzed represented by n=X,X in the category titles.
Time Frame: as for outcome 17
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | GSK2862277 26 mg (BAL Collapsed Lung) | GSK2862277 26 mg (BAL Ventilated Lung)
Number analyzed (Participants) | 8 | 9
Hours
  t1/2, n=0,0: number analyzed (Participants) | 0 | 0
  Tmax, n=3,6: number analyzed (Participants) | 3 | 6
  Tmax, n=3,6 | 7.584 (11.4958) | 7.583 (11.4119)

20. Secondary Outcome: Ratio of Total Protein Derived From BAL and Plasma Values
Description: BAL sampling and plasma sampling was done on Day 1 (on completion of surgery). Raw summary statistics for the derived ratio were not produced. Only statistical modeling was performed that produced a posterior distribution for each treatment. Summary measure for the posterior distribution was the median. The quantity being modeled was the mean treatment effect (pooling data from BAL Collapsed and Ventilated Lungs). The standard deviation is capturing the dispersion of the estimate for the mean effect. Ratio of total protein (Ratio was derived from BAL and Plasma values) is presented.
Time Frame: Day 1 (on completion of surgery)
Population: PP1 Population.
Measure: Median (Standard Deviation); unit: Ratio
Groups:
- Placebo (Pooling BAL Collapsed and Ventilated Lungs): Eligible participants received a single dose of matching placebo on Day 1 via oral inhalation route over approximately 3 to 5 minutes; approximately 1 to 3 hours prior to scheduled surgery. After surgery, participants in this arm underwent either collapsed lung BAL procedure or ventilated lung BAL procedure on Day 1.
- GSK2862277 26 mg (Pooling BAL Collapsed and Ventilated Lungs): Eligible participants received a single dose of GSK2862277 26 mg on Day 1 via oral inhalation route over approximately 3 to 5 minutes; approximately 1 to 3 hours prior to scheduled surgery. After surgery, participants in this arm underwent either collapsed lung BAL procedure or ventilated lung BAL procedure on Day 1.
Arm/Group | Placebo (Pooling BAL Collapsed and Ventilated Lungs) | GSK2862277 26 mg (Pooling BAL Collapsed and Ventilated Lungs)
Number analyzed (Participants) | 15 | 13
Ratio | 0.005 (0.0020) | 0.002 (0.0009)

21. Secondary Outcome: Number of Participants With Positive Immunogenicity Results Post-dosing
Description: Serum samples were obtained to determine incidence and titers of serum anti-GSK2862277 antibodies at the specified time points. The binding antibody detection assay was performed at the specified time points. Number of participants with positive immunogenicity results post-dosing is presented.
Time Frame: Day 8 and Day 31
Population: Safety Population.
Measure: Number; unit: Participants
Arm/Group | Placebo (BAL Collapsed Lung) | Placebo (BAL Ventilated Lung) | GSK2862277 26 mg (BAL Collapsed Lung) | GSK2862277 26 mg (BAL Ventilated Lung)
Number analyzed (Participants) | 5 | 11 | 8 | 9
Participants | 0 | 0 | 0 | 0

22. Secondary Outcome: BAL Concentrations of GSK2862277
Description: BAL samples were collected on Day 1 (on completion of surgery) and BAL concentrations of GSK2862277 and derived PK parameters were determined. Only those participants available at the specified time points were analyzed.
Time Frame: Day 1 (on completion of surgery)
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | GSK2862277 26 mg (BAL Collapsed Lung) | GSK2862277 26 mg (BAL Ventilated Lung)
Number analyzed (Participants) | 1 | 5
Nanograms per milliliter | 11220.00 (NA) — Standard deviation could not calculated as a single participant was analyzed. | 74155.37 (377)

ADVERSE EVENTS:
Time Frame: Serious adverse events and non-serious adverse events were collected from start of the study medication (Day 1) to Follow-up (Day 31)
Description: Serious adverse events and non-serious adverse events were collected for the Safety Population which comprised of all participants who received at least one complete dose of study treatment.
Arm/Group | Placebo (BAL Collapsed Lung) | Placebo (BAL Ventilated Lung) | GSK2862277 26 mg (BAL Collapsed Lung) | GSK2862277 26 mg (BAL Ventilated Lung)
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/11 | 0/8 | 0/9
Serious Adverse Events (participants affected / at risk) | 3/5 | 5/11 | 5/8 | 4/9
Other Adverse Events (participants affected / at risk) | 5/5 | 10/11 | 5/8 | 8/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (BAL Collapsed Lung) (N=5) | Placebo (BAL Ventilated Lung) (N=11) | GSK2862277 26 mg (BAL Collapsed Lung) (N=8) | GSK2862277 26 mg (BAL Ventilated Lung) (N=9)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Splenic infarction (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diaphragmatic hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal ischaemia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Complication associated with device (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Empyema (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2) | 2 (3) | 1 (1)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Failure to anastomose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anastomotic leak (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Iatrogenic injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Procedural pneumothorax (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Diaphragmatic rupture (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Femoral artery embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (BAL Collapsed Lung) (N=5) | Placebo (BAL Ventilated Lung) (N=11) | GSK2862277 26 mg (BAL Collapsed Lung) (N=8) | GSK2862277 26 mg (BAL Ventilated Lung) (N=9)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Anaemia folate deficiency (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 2 (2) | 1 (1) | 1 (2)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Diabetic retinopathy (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Visual acuity reduced (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypothermia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 3 (3) | 2 (3) | 1 (1)
Catheter site haemorrhage (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Catheter site haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Catheter site discharge (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Complication associated with device (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pneumonia klebsiella (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Febrile infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Enterobacter sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wound infection staphylococcal (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Klebsiella infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infectious pleural effusion (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stoma site cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anaemia postoperative (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Postoperative hernia (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Procedural hypotension (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Endotracheal intubation complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Unintentional medical device removal (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2) | 2 (2) | 2 (2) | 2 (2)
Blood albumin decreased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Blood calcium decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood lactic acid increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood sodium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood urea increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Electrocardiogram T wave inversion (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Glomerular filtration rate decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematocrit decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Monocyte count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Oxygen saturation decreased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PO2 decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Red blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Reticulocyte count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Blood phosphorus decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Platelet count increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Nasogastric output high (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fungal test positive (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 4 (4) | 1 (1) | 0 (0)
Urine output decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram change (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Staphylococcus test positive (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Streptococcus test positive (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Escherichia test positive (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Klebsiella test positive (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Nuclear magnetic resonance imaging spinal abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Magnesium deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mineral deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 2 (2)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dizziness postural (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urine odour abnormal (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (4) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2016-08-23): https://cdn.clinicaltrials.gov/large-docs/37/NCT02221037/Prot_000.pdf
  • Statistical Analysis Plan (2015-11-17): https://cdn.clinicaltrials.gov/large-docs/37/NCT02221037/SAP_001.pdf